CLINICAL TRIAL: NCT00150137
Title: The Influence of Continuous Treatment With Antithyroid Drugs on the Effect of Radioiodine in Patients With Hyperthyroidism
Brief Title: Antithyroid Drugs During Radioiodine Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 013
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-02-03 (Estimated); Status verified 2005-09

CONDITIONS: Toxic Nodular Goitre; Graves Disease
Keywords: Radioiodine therapy; Graves' disease; toxic nodular goiter; antithyroid drugs; radioprotection
MeSH Terms: conditions — Graves Disease | interventions — Methimazole

INTERVENTIONS:
Drug: Methimazole

SUMMARY:
Background: The use of radioactive iodine (131I) therapy as the definite cure of hyperthyroidism is widespread. According to a survey on the management of Graves' disease, thirty per cent of physicians prefer to render their patients euthyroid by antithyroid drugs (ATD) prior to 131I therapy. This strategy is presumably chosen to avoid 131I induced 'thyroid storm', which, however, is rarely encountered. Several studies have consistently shown that patients who are treated with ATD prior to 131I therapy have an increased risk of treatment failure. Mostly, patients with Graves' disease have been studied, while other studies were addressed also toxic nodular goiter. Thus, it is generally accepted that ATD have 'radioprotective' properties, although this view is almost exclusively based on retrospective data and is still under debate (13). Indeed, this dogma was recently challenged by two randomized trials in Graves' disease, none of which showed such an adverse effect of methimazole pretreatment. It cannot be excluded that the earlier results may have been under influence of selection bias, a source of error almost unavoidable in retrospective studies. Whether ATD is radioprotective also when used in the post 131I period has also been debated. In the early period 131I therapy following a transient rise in the thyroid hormones is seen which may give rise to discomfort in some patients. The continuous use of ATD during 131I therapy leads to more stable levels of the thyroid hormones. By resuming ATD following 131I therapy, euthyroidism can usually be maintained until the destructive effect of 131I ensues. Nevertheless, many physicians prefer not to resume ATD, probably due to reports supporting that such a strategy reduces the cure rate. Parallel to the issue of ATD pretreatment, the evidence is based on retrospective studies and the ideal set-up should be reconsidered. To underscore the importance of performing randomized trials we showed recently that resumption of methimazole seven days after 131I therapy had no influence on the final outcome.

Aim: To clarify by a randomized trial whether continuous use of methimazole during radioiodine therapy influences the final outcome of this therapy, in a comparison with a regime in which methimazole as mono-therapy is discontinued 8 days before radioiodine.

Patients and Methods: 80 consecutive patients suffering from recurrent Graves' disease or a toxic nodular goiter are included. All patients are rendered euthyroid by methimazole (MMI) and randomized either to stop MMI eight days before 131I or to continue MMI until four weeks after 131I. Calculation of the 131I activity (max. 600 MBq) includes an assessment of the 131I half-life and the thyroid volume. Patients are followed for one year with close monitoring of the thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* Hyperthyroid patients going to be treated with radioiodine either due to recurrent Graves' disease or toxic nodular goiter.

Exclusion Criteria:

* Age < 18 yrs.
* Allergy to anti-thyroid drugs
* Substernal or large (> 100ml) goiter
* Severe endocrine ophthalmopathy
* Pregnancy or lactation
* Suspicion of thyroid malignancy
* Unsafe contraconception
* Physical or mental condition that hinders corporation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Thyroid function after one year of follow-up

SECONDARY OUTCOMES:
Thyroid radioiodine 131I uptake
Thyroid volume after one year of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Steen J Bonnema, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark